CLINICAL TRIAL: NCT03323021
Title: A Single-Center Double Arm Single-Blinded Randomized Screening Clinical Trial to Evaluate the Use of Human Dehydrated Amnion/Chorion Membrane to Facilitate the Recovery of Renal Function Following Robotic Partial Nephrectomy
Brief Title: Use of Human Dehydrated Amnion/Chorion (DHACM) Allograft in Partial Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFSUR001
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Partial Nephrectomy; Kidney Cancer; Renal Function Aggravated
MeSH Terms: conditions — Kidney Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with DHACM (Experimental): Partial nephrectomy patched with DHACM
  Interventions: Other: Dehydrated human amnion/chorion membrane
- Control without DHACM (Active Comparator): Partial nephrectomy without DHACM.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Dehydrated human amnion/chorion membrane — dehydrated human amnion/chorion membrane
  Arms: Treatment with DHACM
Other: Standard of Care — Standard of Care
  Arms: Control without DHACM

SUMMARY:
After partial nephrectomy, kidney function decreases by about 10% overall and by about 20% in the operated kidney. This is primarily due to the loss of healthy parenchymal volume during resection of the tumor. In an effort to preserve and regenerate healthy parenchyma during the procedure and ultimately renal function after partial nephrectomy, the single center double arm single-blinded randomized screening clinical trial will evaluate the ability of human amnion/chorion allograft to facilitate the recovery of renal function following robotic partial nephrectomy.

DETAILED DESCRIPTION:
To determine whether Amniofix facilitates improved recovery of renal function at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Any individual with a diagnosis of a renal mass.
* All Patients undergoing partial nephrectomy as their definitive treatment for their renal mass.
* Ability to understand and the willingness to sign a written informed consent.
* Patients with a solitary clinical T1a renal mass.

Exclusion Criteria:

* Patients undergoing radical nephrectomy as their definitive treatment for their renal mass.
* Patients with Transitional Cell Carcinoma.
* Patients with known hereditary syndromes such Von Hippel-Lindau (VHL) syndrome, Lynch Syndrome, Birt-Hogg-Dube Syndrome.
* Patients with metastatic disease undergoing cytoreductive nephrectomy as their definitive treatment for metastatic disease.
* Patients with prior kidney surgery.
* Patients with a solitary or horseshoe kidney.
* Patients with a positive margin found during intra-operative frozen section done only when clinically indicated (i.e., macroscopic abnormality identified).
* Patients with multiple renal masses.
* Patients with greater than a clinical T1a renal mass.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
Recovery of Renal Function | 12 months
  Evaluation of GlomerularFiltration Rate (GFR)

SECONDARY OUTCOMES:
Preservation of Renal Parenchymal Volume | 12 months
  Using radiologic computed tomography measurements
Cancer Control Rates | 12 months
  Observed recurrence rate

CONTACTS AND LOCATIONS:
Overall Officials: Ketan Badani, MD, Principal Investigator — Mt. Sinai Medical Center
Locations (1):
- The Mount Sinai Hospital, New York, New York, United States